CLINICAL TRIAL: NCT00103233
Title: A Randomized Study of Weekly Vinorelbine (Navelbine®) Alone or in Combination With Trastuzumab (Herceptin®) (NSC-688097) for Patients With HER-2-Positive Metastatic Breast Cancer Whose Tumors Have Progressed After Taxane + Trastuzumab Combination Therapy - Phase III
Brief Title: Vinorelbine With or Without Trastuzumab in Treating Women With Progressive Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000409573; SWOG-S0347
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2005-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Vinorelbine

INTERVENTIONS:
Biological: trastuzumab
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Trastuzumab may also help vinorelbine work better by making tumor cells more sensitive to the drug. Giving vinorelbine together with trastuzumab may be an effective treatment for breast cancer. It is not yet known whether giving vinorelbine together with trastuzumab is more effective than vinorelbine alone in treating breast cancer.

PURPOSE: This randomized phase III trial is studying vinorelbine and trastuzumab to see how well they work compared to vinorelbine alone in treating women with progressive metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare progression-free survival (PFS) of women with HER2-positive progressive metastatic breast cancer treated with vinorelbine with or without trastuzumab (Herceptin®).
* Compare overall survival and time to treatment failure in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the response rate (complete and partial, confirmed and unconfirmed) in patients with measurable disease treated with these regimens.
* Correlate baseline circulating tumor cells (CTC) with PFS, overall survival, and disease progression status at 9 weeks in patients treated with these regimens.
* Correlate 4-week CTC with subsequent PFS and overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive trastuzumab (Herceptin®) IV over 90 minutes and vinorelbine IV over 10 minutes on day 1 of course 1. Patients receive trastuzumab IV over 30 minutes and vinorelbine IV over 10 minutes on days 1, 8, 15, and 22 in all subsequent courses. If trastuzumab is discontinued due to toxicity, patients may continue to receive vinorelbine alone.
* Arm II: Patients receive vinorelbine IV over 10 minutes on days 1, 8, 15, and 22.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 292 patients (146 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Clinical evidence of metastatic disease
* HER2-positive tumor, as indicated by one of the following methods:

  * HER2 gene amplification by fluorescence in situ hybridization
  * HER2 protein overexpression (3+) by immunohistochemistry
* Disease progression during or after prior taxane therapy (single-agent paclitaxel, docetaxel, or taxane-containing combination chemotherapy) in combination with trastuzumab (Herceptin®) as first- or second-line chemotherapy for metastatic disease

  * Patients who received maintenance therapy with single-agent trastuzumab after acheiving a response or stable disease to prior taxane/trastuzumab combination therapy are eligible provided disease has progressed
* Measurable or nonmeasurable disease

  * No effusions or ascites as the only sites of disease
* No leptomeningeal disease or lymphatic pulmonary metastases
* Brain metastases allowed provided disease is stable for > 3 months after completion of prior radiotherapy to the brain
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* SGOT or SGPT ≤ 2.5 times upper limit of normal (ULN) (< 5 times ULN in the presence of liver metastases)
* Alkaline phosphatase ≤ 3 times ULN (< 5 times ULN in the presence of liver or bone metastases)

Renal

* Creatinine ≤ 2.0 mg/dL
* Calcium ≤ 11.0 mg/dL

Cardiovascular

* No history of significant symptomatic cardiac disease
* LVEF ≥ 50% of the lower limit of normal by MUGA or ECG

Other

* No pre-existing clinically significant (≥ grade 2) motor or sensory neuropathy except for abnormalities due to cancer
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 28 days since prior trastuzumab
* No concurrent filgrastim (G-CSF)

Chemotherapy

* See Disease Characteristics
* No more than 2 prior chemotherapy regimens for metastatic breast cancer

  * Prior adjuvant/neoadjuvant chemotherapy allowed, for a total of 3 prior regimens
* No prior vinorelbine
* No other prior chemotherapy after progression on a taxane/trastuzumab regimen
* No prior cumulative dose > 360 mg/m^2 of anthracycline-based chemotherapy

Endocrine therapy

* No prior hormonal therapy after progression on a taxane/trastuzumab regimen
* Prior exogenous hormonal therapy for stage IV disease and/or as adjuvant therapy allowed

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to > 50% of the marrow-bearing bone

Surgery

* At least 4 weeks since prior major surgery (2 weeks for minor surgery) and recovered

Other

* Concurrent bisphosphonates allowed for bone metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, MD, MPH, DPhil — M.D. Anderson Cancer Center; Francisco J. Esteva, MD — M.D. Anderson Cancer Center